CLINICAL TRIAL: NCT07318376
Title: Effect of E-learning Training on National Institutes of Health Stroke Scale (NIHSS) and Modified Rankin Scale (mRS) Assessment Performance: a Web-based Randomized Controlled Trial
Brief Title: Effect of E-learning Training on National Institutes of Health Stroke Scale (NIHSS) and Modified Rankin Scale (mRS) Assessment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stuby Loric (Other)
Collaborators: University Hospital, Geneva (Other); Geneve TEAM Ambulances (Other)
Responsible Party: Sponsor-Investigator, Stuby Loric, Principal Investigator, Geneve TEAM Ambulances
Organization: Geneve TEAM Ambulances (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NIHSS-6
Record Dates: First submitted 2025-12-23; First posted 2026-01-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Stroke Assessment; National Institutes of Health Stroke Scale; Modified Rankin Scale; Clinical Competence; Education; Distance Learning-Online Learning
Keywords: E-learning; Web-based training; Stroke assessment; National Institutes of Health Stroke Scale (NIHSS); Modified Rankin Scale (mRS); Paramedics; Emergency Medical Services; Prehospital care; Clinical competence; Educational intervention; Randomized controlled trial; Performance assessment; Distance education; Continuing professional education
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Control group: Participants will first complete the NIHSS quiz and mRS case vignettes without prior training.
- Intervention group (Experimental): Participants will follow the e-learning modules (NIHSS and mRS).
  Interventions: Other: Educational intervention

INTERVENTIONS:
Other: Educational intervention — Educational intervention by the mean of an e-learning modules (NIHSS and mRS).
  Arms: Intervention group

SUMMARY:
The goal of this web-based randomized clinical trial is to evaluate whether an e-learning training program improves the accuracy of National Institutes of Health Stroke Scale (NIHSS) and modified Rankin Scale (mRS) assessments among practicing paramedics in French-speaking Switzerland who have not previously received formal training in these scales.

The main questions it aims to answer are:

* Does e-learning training improve performance on a standardized NIHSS assessment quiz compared with no prior training?
* Does e-learning training improve the accuracy of mRS assessment using case-based clinical vignettes compared with no prior training?

Researchers will compare paramedics who complete the NIHSS and mRS e-learning modules before assessment (intervention group) with paramedics who complete the assessments without prior training (control group) to determine whether e-learning training leads to higher assessment performance scores.

Participants will:

* Provide electronic informed consent via a secure web-based platform
* Be randomly assigned to either the intervention group or the control group
* Complete either the e-learning modules before assessment or the assessments before training, depending on group allocation
* Complete an online NIHSS quiz and mRS case-based vignettes
* Receive access to the NIHSS and mRS e-learning modules by the end of the study

ELIGIBILITY:
Inclusion Criteria:

* Holding a paramedic title (recognized in Switzerland)
* Currently actively practicing in Switzerland
* Fluent in French (all study material will be provided in French)

Exclusion Criteria:

* Previously completed formal training on either the NIHSS or the mRS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Performance on a NIHSS 50-item quiz | From enrollment to the end of the study path in a timeframe of maximum 4 weeks.
  The primary outcome will be the performance on a NIHSS 50-item quiz consisting in 3 full assessments of a patient (3x15 items) plus 5 general questions (each question scores 1 point if correct, maximum total of 50 points).

SECONDARY OUTCOMES:
Performance of mRS assessment | From enrollment to the end of the study path in a timeframe of maximum 4 weeks.
  The secondary outcome will be the performance of mRS assessment of about 10 newly developed case-based vignettes (each question scores 1 point if correct, maximum total of 10 points).

CONTACTS AND LOCATIONS:
Overall Officials: Loric Stuby, Principal Investigator — Genève TEAM Ambulances
Locations (1):
- Genève TEAM Ambulances, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Study data will be made available by deposition in a public repository (Yareta.org).